CLINICAL TRIAL: NCT01966185
Title: Establishing Learning Curves in Virtual Simulation Training of Mastoidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Steven Andersen, Research fellow, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: H-4-2013-FSP-088
Record Dates: First submitted 2013-10-11; First posted 2013-10-21 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: User-Computer Interface; Clinical Skills; Motor Skills; Temporal Bone; Students
Keywords: virtual simulation; temporal bone; surgical training; medical education; self-directed learning; final product assessment; cognitive load; reaction time; skills training; simulator metrics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tutor function off (No Intervention): The tutor function will be off for 12 out of 12 repeat simulations.
- Tutor function on (Experimental): The group will have the tutor function on for the 5 first out of 12 repeat simulation sessions.
  Interventions: Other: Tutor function on

INTERVENTIONS:
Other: Tutor function on — The simulator-integrated tutor function with volumetric green lighting of the intended volume to be drilled.
  Arms: Tutor function on

SUMMARY:
The purpose of this study is to establish learning curves of mastoidectomy training in virtual surgical simulation training, to establish the long-term effect of repeat simulation training and to explore the transfer of skills, the roles of an integrated tutor function, self-directed learning and cognitive load.

DETAILED DESCRIPTION:
Repeat surgical simulation training is known to provide better learning and long-term transfer. The learning curves for the mastoidectomy procedure have not been intensively studied. The only study conducted on learning curves in mastoidectomy to date found a plateau in performance for 4 medical students after about 4 mastoidectomy procedures on separate occasions. The participants were however assessed using an unvalidated, unestablished simulator integrated overall performance score. There is therefore a need for establishing learning curves and plateau using established objective assessment scales, which could have implications for future studies and on a larger scale for the future organization of temporal bone dissection courses.

The long-term effect on learning of deliberate repeat simulator training of the mastoidectomy procedure has not previously been studied. The role of cognitive load in learning complex surgical technical skills in simulation has not been studied in great detail. The relationship between time and progress/performance assessment using Final Product Analysis (FPA) has not been studied.

We have previously suggested that a tutor-function with volumetric approach with green lighting of the procedural steps could have an effect on performance. The effect of the tutor function could however not be isolated.

ELIGIBILITY:
Inclusion Criteria:

* medical students
* informed written consent

Exclusion Criteria:

* prior training on the Visible Ear Simulator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in Final Product Assessment Score | 4 months
  Mastoidectomy final product assessment score using a modified Welling Scale for performance assessment.

SECONDARY OUTCOMES:
Change in simulator metrics | 4 months
  Integrated simulator metrics on volume drilled (inside+outside target volumes), collisions with vital structures in simulation, time.
Change in reaction time | 4 months
  Reaction time to a visual cue (in ms)

OTHER OUTCOMES:
Background data | At recruitment
  Background data from a questionnaire including questions on demographics, prior simulation training and experience and interests in computers and IT

CONTACTS AND LOCATIONS:
Overall Officials: Steven AW Andersen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark